CLINICAL TRIAL: NCT01725932
Title: A Multicentre Randomised Controlled Trial of Culturally Adapted CBT Based Self Help Manual for Depression in Pakistan
Brief Title: Randomized Controlled Trial of Cognitive Therapy Based Self Help Manual for Depression
Acronym: CaCBT_SH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACT_SHCBTD_2012
Record Dates: First submitted 2012-10-31; First posted 2012-11-14 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: culture, depression, cognitive therapy, behaviour therapy,
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Culturally adapted CBT based Self Help (Experimental): Culturally sensitive cbt based self help intervention, which consists of 6 regular chapters and 2 additional chapters. The self help intervention involves family to improve compliance with the intervention
  Interventions: Behavioral: Culturally adapted CBT based Self Help
- Care As Usual (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Culturally adapted CBT based Self Help — Intervention was based on our initial work using mixed methods, using mixed methods,in Pakistan. It focused on psycho-education, symptoms management, changing negative thinking, behavioral activation, problem solving, improving relationships and communication skills. One person from the family was involved in all cases. The intervention consists of 7 chapters. Manual can be used by the patient's or carers with at least 5 years of education. A member of the research team called them once every week to remind them of the next chapter and also to discuss any issues o problems that emerged during the previous week. This manual can be downloaded from PACT website (http://www.pactorganization.com/)
  Arms: Culturally adapted CBT based Self Help

SUMMARY:
While CBT (Cognitive Behaviour Therapy)has been found to be effective in treating depression in West, only limited amount of research has been conducted to find assess its effectiveness in low and middle income countries. We have developed culturally sensitive CBT during the last few years in Pakistan. Pakistan has high rates of depression. And there is currently a need to develop and test evidence based treatments which are culturally sensitive and cost effective. IN this project we will be assessing the effectiveness of a culturally sensitive CBT based self help intervention for depression in Pakistan against care as usual, using a randomized controlled design.

ELIGIBILITY:
Inclusion Criteria:

* All those who fulfil the diagnosis of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4 ) using ICD10 RDC (International Classification of Diseases, Research Diagnostic Criteria), scored 8 or more on HADS (Hospital Anxiety and Depression Scale) Depression Sub-scale, are between the ages of 18-60 and either patient or the carer has at least 5 years of education.

Exclusion Criteria:

* The exclusion criteria include; excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence) significant cognitive impairment (for example learning disability or dementia) and active psychosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and depression Rating Scale- Depression subscale | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of depression

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale, Anxiety subscale | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of anxiety
Bradford Somatic Inventory | Participants will be assessed at baseline and then end of therapy at 12 weeks
  Measurement of somatic symptoms
Brief disability questionnaire | Participants will be assessed at baseline and then end of therapy at 12 weeks
  To measure disability associated with depression

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Khalid, MSc, Study Director — PACT